CLINICAL TRIAL: NCT04215783
Title: Childhood Allergy and the Neonatal Environment
Acronym: CANOE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1103; 5UH3OD023282 (NIH); 1U24AI152177-01 (NIH); MSN236000 (Other Grant/Funding Number: NIH ECHO program); A536770 (Other: UW Madison); SMPH/PEDIATRICS/AIR (Other: UW Madison); Protocol Version 1/23/2026 (Other: UW Madison)
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Asthma in Children; Allergy
Keywords: Allergy, Asthma, Children, Birth cohort
MeSH Terms: conditions — Hypersensitivity; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cryopreserved samples of serum, plasma, urine, and nasal secretions or wash fluid, will be analyzed for proteins or metabolites that may serve as biomarkers for exposures or for study outcomes. A genetic sample (blood buffy coat or saliva) from the mother and child will be saved (if they agree) for use later to look at DNA, RNA or both.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research study is to study the relationship between childhood asthma, allergies, and early-life environmental factors that may cause childhood asthma and allergies. Previous birth cohort studies have found early-life environmental factors such as allergies, pollutants, viruses and bacteria have all contributed to the development of asthma and allergies. Investigators are doing this research because there continues to be a strong need to understand the root causes of asthma and allergies. The CANOE study is an observational cohort study, which means investigators are not asking participants or participant's child to change their medications and investigators will not be giving participants or participant's child a study drug.

DETAILED DESCRIPTION:
The CANOE study will provide an opportunity to collect novel longitudinal samples not available from the current CANOE birth cohorts, as well as enhanced and standardized environmental sampling in early life. One of the main goals of this study is to gather data and specimens, beginning in the prenatal periods, that will assess environmental exposures to toxins and microbes, and host characteristics including genetics, epigenetics, gene expression, the proteome and metabolome, microbial colonization and viral respiratory infections. The main study outcomes will be important interim conditions (e.g., recurrent wheeze, early multiple sensitization) that are highly associated with the development of asthma. Additional outcomes (perinatal outcomes, growth, neurocognitive development) will be collected as part of the collaborative Environmental Influences on Child Health Outcomes (ECHO)-wide Cohort Data Collection Protocol.

ELIGIBILITY:
Inclusion Criteria:

1. History of or concurrent asthma or allergic rhinitis (hay fever) in either biologic parent or sibling (at least one shared biological parent) by parental report. The presence of paternal or sibling allergy or asthma will be ascertained by maternal report.
2. Maternal age greater than or equal to 18 years at the time of study enrollment.

Exclusion Criteria:

1. Maternal HIV infection at time of delivery.
2. Plans for the family to move out of the geographic area during the period of the study.
3. Does not speak English.
4. Current maternal use of progesterone during pregnancy to prevent preterm birth.

   * Progesterone use is only an exclusion if currently being taken at time of enrollment for preterm birth. Previous use to prevent preterm birth or use at any time for other indications is allowed.
5. Pregnancy is a result of an embryo donor (egg and sperm donor pregnancies are permitted).
6. Past or current medical problems or findings from physical examination or laboratory testing which, in the opinion of the investigator or designee, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study participants of CANOE will consist of four ethnically diverse cohorts from predominantly urban and suburban families at 4 sites. Previous studies have identified common themes in populations of children who differ by ethnicity and environmental exposures. These include inverse relationships between wheezing and/or atopy and exposure to specific microbes and allergens in early life. Obtaining prospective data from newly recruited participants during the prenatal period offers multiple opportunities to optimize sample collection for assessment of environmental exposures and enhance the scientific value of the CREW consortium. To enrich the cohort for the development of wheezing and allergic sensitization, we will enroll participants with a family history of asthma or allergies.
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of children with recurrent wheeze | 3 years
  Number of children with recurrent wheezing will be reported. Recurrent wheeze, defined as at least 2 episodes of wheeze with one occurring in the last 12 months of study participation for children between 2 and 3 years of age.
Number of children with early aeroallergen sensitization | 2 years
  Number of children with early aeroallergen sensitization will be reported. Early aeroallergen sensitization, defined as sensitization to at least one aeroallergens by age 2 years.
Number of children diagnosed with asthma | 4 years
  Number of children who diagnosed, either by a doctor or self-report, at age 6 or 7 years.

SECONDARY OUTCOMES:
Number of children with Atopic dermatitis (AD) | 3 years
  Number of children with AD will be reported. Atopic dermatitis, defined if at least 1 of the following is present:
  1. Physician diagnosis of eczema/AD (either study physician or other physician by parental report) at any time,
  2. Objective SCORAD (SCORing Atopic Dermatitis) ≥ 8 at 1 or more study assessments. The range of the objective SCORAD lies between 0 and 83. Based on the objective SCORAD, the severity of AD can be classified into mild (<15), moderate (between 15 and 40) and severe (greater than or equal to 40) AD.
  3. Parent report of an itchy rash outside of the diaper area lasting for at least 7 days and not diagnosed as another condition.
Number of children with food allergies | 3 years
  Number of children with the food allergy will be reported. Food allergy defined as typical signs and symptoms of immediate IgE (Immunoglobulin E) -mediated reaction (such as urticaria, angioedema, vomiting, wheezing, cough, hypotension) within 2 hours of food ingestion and with positive immunocap testing to that food.
Lung function | 4 years
  Lung function is assessed by spirometry, a 10-15 minute, non-invasive, and painless test that requires participants to breathe through a mouthpiece connected to a computer, often with a nose clip to prevent air leaks. Spirometry measures lung function by calculating the volume and speed of air exhaled, and is reported as a ratio of the two.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Singh, MD, Principal Investigator — UW Madison; James Gern, MD, Principal Investigator — UW Madison
Locations (4):
- United States (4):
  - Henry Ford Health Systems, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No